CLINICAL TRIAL: NCT02109406
Title: A Randomized, Double Blind, Chronic Dosing (14 Days), Three Period, Placebo Controlled, Cross Over, Multi Center Study to Assess Efficacy and Safety of Two Dose Levels of AZD2115 MDI in Subjects With Moderate to Severe COPD
Brief Title: Efficacy and Safety Study of Two Dose Levels of AZD2115 in Subjects With Moderate to Severe COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZD2115 D3060C00006
Record Dates: First submitted 2014-04-02; First posted 2014-04-09 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD2115 Dose 1 (Experimental): AZD 2115, Dose 1 administered as two inhalations BID
  Interventions: Drug: AZD2115 Dose 1
- AZD 2115 Dose 2 (Experimental): AZD 2115, Dose 2 administered as two inhalations BID
  Interventions: Drug: AZD 2115, Dose 2
- Placebo MDI (Placebo Comparator): Placebo MDI administered as two inhalations BID
  Interventions: Drug: Placebo MDI

INTERVENTIONS:
Drug: AZD2115 Dose 1 — AZD 2115, Dose 1 administered as two inhalations BID
  Arms: AZD2115 Dose 1
Drug: AZD 2115, Dose 2 — AZD 2115, Dose 2 administered as two inhalations BID
  Arms: AZD 2115 Dose 2
Drug: Placebo MDI — Placebo MDI administered as two inhalations BID
  Arms: Placebo MDI

SUMMARY:
This is a phase IIa dose-ranging, randomized, double-blind, chronic-dosing (14 Days), three-period, placebo-controlled, multi-center, cross-over study to assess the efficacy and safety of two dose levels of a dual pharmacology molecule with the combined properties of a long-acting muscarinic antagonist (LAMA) and a long-acting beta-agonist (LABA); (AZD2115) delivered by a metered-dose inhaler (MDI) in subjects with moderate to severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease Diagnosis: Subjects with an established clinical history of COPD for more than 1 year at Screening, according to the COPD GOLD guidelines.
* Current or former smokers with a history of ≥10 pack years of cigarette smoking.
* Post-bronchodilator FEV1/FVC ratio of <70%.
* Pre-bronchodilator FEV1 must be <80% predicted
* Women of non-child bearing potential (ie., physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal); or women of child bearing potential, has a negative serum pregnancy test at Screening and agrees to acceptable contraceptive methods for the duration of the study.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating.
* Significant diseases other than COPD, ie., disease or condition which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study.
* Primary diagnosis of asthma.
* Alpha-1 antitrypsin deficiency as the cause of COPD
* Other active pulmonary disease such as active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, idiopathic interstitial pulmonary fibrosis, primary pulmonary hypertension, or uncontrolled sleep apnea.
* Poorly controlled COPD (hospitalization due to poorly controlled COPD within 3 months of Screening or requiring treatment with corticosteroids or antibiotics in the 6 week interval prior to Screening or during Screening.
* Unstable ischemic heart disease, left ventricular failure, or documented myocardial infarction within 12 months of Randomization.
* Clinically significant abnormal ECG.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) area under the curve from 0 to 12 hours (AUC0-12) relative to baseline | 14 Days

SECONDARY OUTCOMES:
Change from baseline in morning pre dose trough FEV1 | 14 Days
Peak change in FEV1 | 14 Days
Forced vital capacity (FVC) AUC0-12 relative to baseline | 14 Days
Peak change in FEV1 | Day 1
Change from baseline in 12-hour post dose trough FEV1 | 14 Days
Time to onset of action | Day 1

OTHER OUTCOMES:
Pharmacokinetics | Day 1 through Day 15
  Cmax, AUC0-12, AUC0-t, tmax, Apparent elimination half-life (t1/2), Apparent volume of distribution (Vd/F), Apparent total body clearance (CL/F)
Safety | Day1 through Day 15
  Safety will be assessed by adverse events (AEs), physical examination findings, dry mouth and tremor assessments, paradoxical bronchospasm, vital signs, electrocardiogram (ECG), and laboratory assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Siddiqui, MD, Study Director — Pearl Therapeutics, Inc.
Locations (3):
- United States (3):
  - Pearl Therapeutics Study Site, Clearwater, Florida
  - Pearl Therapeutics Study Site, Charleston, South Carolina
  - Pearl Therapeutics Study Site, Spartanburg, South Carolina